CLINICAL TRIAL: NCT03526445
Title: Hepatic Metabolic Changes in Response to Glucagon Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18003696
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Total Pancreatectomy; Diabetes Mellitus
Keywords: Glucagon; Stable isotope; Energy expenditure; Lipid metabolism; Glucose metabolism; Appetite
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus | interventions — Glucagon; Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucagon (Active Comparator): 3 hours i.v. infusion of Glucagon (4 ng/kg/min).
  Interventions: Drug: Glucagon
- Saline (Placebo Comparator): 3 hours i.v. infusion of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Glucagon — Glucagon (4 ng/kg/min)
  Other Names: GlucaGen
  Arms: Glucagon
Drug: Saline — Placebo
  Arms: Saline

SUMMARY:
The objective of the study is to investigate how exogenously administered glucagon affects hepatic lipid, glucose and protein metabolism as well as appetite, food intake and resting energy expenditure.

DETAILED DESCRIPTION:
Most research has focused on the role of the pancreatic hormone, insulin, and insulin signalling (or lack of) in the development of NAFLD. However, increasing evidence suggest that the other major gluco-regulatory pancreatic hormone glucagon is also implicated in lipid metabolism and recent human data from studies investigating the effect of glucagon receptor antagonism suggest that glucagon signalling may be essential for maintaining a fat-free liver. This, combined with observations of increased degree of hepatic steatosis in patients after total pancreatectomy, who are devoid of pancreatic glucagon and typically are lean and peripherally insulin sensitive, suggests that glucagon may play a hitherto unrecognised role in the pathophysiology of NAFLD.

The hypothesis of the study is that exogenously delivered glucagon will drive hepatic metabolism in a lipolytic direction and increase resting energy expenditure without affecting appetite and food intake.

The acute effects of exogeneous glucagon infusion on hepatic lipid metabolism will be evaluated in patients after total pancreatectomy (no endogenous pancreatic hormones), in patients with type 1 diabetes (no endogenous insulin production) and in healthy controls (preserved endogenous pancreatic hormones).

ELIGIBILITY:
Inclusion Criteria:

Pancreatectomised patients

* Patients who have undergone total pancreatectomy
* Caucasian between 30-80
* Blood haemoglobin >7.0 mmol/l for males and >6.5 mmol/l for females
* Informed consent

Patients with type 1 diabetes

* Patients with C-peptide negative type 1 diabetes
* Caucasian between 30-80
* Blood haemoglobin >7.0 mmol/l for males and >6.5 mmol/l for females
* Informed consent

Healthy controls

* Normal fasting plasma glucose (< 7 mmol/l) and normal HbA1c (< 6.5 %) (30,31)
* Normal blood haemoglobin (>8.3 mmol/l for males and >7.3 mmol/l for females)
* Caucasian between 30-80
* Informed consent

Exclusion Criteria:

All subjects

* Inflammatory bowel disease
* Gastrointestinal resection (other than the gastro-duodenectomy performed in connection with total pancreatectomy) and/or ostomy
* Nephropathy (eGFR < 60 ml/min/1.73 m² and/or urine albumin > 20 mg/L)
* Known liver disease (excluding non-alcoholic fatty liver disease)
* Severe lung disease
* Pregnancy and/or breastfeeding
* Uncontrolled hypertension and/or significant cardiovascular disease
* Treatment with drugs with potential steatogenic side-effects within three months prior to inclusion
* Alcohol consumption above 21 units/week for men and 14 units/week for women
* Any condition that the investigator feels would interfere with the safety of the trial participation or the safety of the subject.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Hepatic lipid metabolism | -120,-30,-15,0,30,60,90,120,135,150 minutes
  evaluated using isotopic labelled tracer kinetics: lipolysis, ketogenesis, very low-density lipoprotein (VLDL) secretion and free fatty acid (FFA) re-esterification rate

SECONDARY OUTCOMES:
Changes in plasma concentration of lipids | 0, 60,150 minutes
  Total cholesterol, VLDL, LDL, HDL, FFA
Changes in plasma concentration of amino acids | 0, 60, 120, 150 minutes
Changes in plasma concentration of fibroblast growth factor 21 (FGF-21) | -120,0,150 minutes
Endogenous glucose production | -120,-30,-15,0,30,60,90,120,135,150 minutes
  Measured by glucose tracer
Changes in resting energy expenditure and oxidation rate | 0, 150 minutes
  Measured by indirect calorimetry
Food intake | 30 minutes (150-180) minutes
  Ad libitum meal
Changes in appetite sensation | 0,30,60,90,120,150 minutes
  Visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Filip Krag Knop, Prof., Study Director — Center for Clinical Metabolic Research, Gentofte Hospital, University of Copenhagen
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, University of Copenhagen, Hellerup, Denmark